CLINICAL TRIAL: NCT03746912
Title: An Open-Label, Multi-Center, Expanded Treatment Protocol of Quizartinib in Adult Subjects With Relapsed or Refractory Acute Myeloid Leukemia (AML) With FLT3-ITD Mutations
Brief Title: Expanded Treatment Protocol for Adults With FLT3-ITD Mutated Relapsed or Refractory Acute Myeloid Leukemia (AML) to Receive Quizartinib
Status: No longer available | Type: Expanded Access
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: AC220-A-U203
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia With Gene Mutations
Keywords: Refractory or Relapsed; FLT3- internal tandem duplication (ITD) mutation; FLT3-ITD mutation
MeSH Terms: conditions — Recurrence | interventions — quizartinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Quizartinib Dihydrochloride — Tablets for once daily oral administration at doctor-recommended dose in continuous 28-day cycles
  Other Names: Quizartinib

SUMMARY:
An expanded access program (EAP):

* Allows doctors to give medicine to patients,
* Before it is approved by health authorities.

This EAP is for:

* Quizartinib
* Patients with FLT3-ITD mutated AML,
* AML that has come back, or
* Is resistant to other therapies.

A participant will receive quizartinib if:

* The doctor submits a request,
* The participant is eligible, and
* The country allows the EAP.

DETAILED DESCRIPTION:
This is an expanded access program (EAP) providing access to quizartinib for participants with Relapsed/Refractory FLT3-ITD mutated AML, prior to approval by local regulatory agencies. Availability of the EAP is dependent upon physician request, country eligibility and local/country regulations. EAP countries included Austria, Belgium, Brazil, Denmark, France, Germany, Ireland, Italy, Netherlands, Norway, South Korea, Spain, Sweden, Switzerland, Taiwan, Thailand, United Kingdom, and United States. Physicians may request access to the EAP for participants who they feel may benefit from quizartinib and meet the eligibility criteria.

Participants may continue quizartinib until there is a lack of clinical benefit or the occurrence of unacceptable toxicity. Treatment should be interrupted for allogeneic hematopoietic stem cell transplantation (HSCT), but may be resumed after the transplant.

Participant enrollment may continue until 18 months after regulatory approval, depending on country regulation; or until such time the marketed medication is available, whichever occurs first.

Participants will be asked to follow the care as outlined by their treating physician. Participants will be followed for 30 days after their final treatment or until the patient is transitioned to commercially available product. Physicians will be required to report safety data to Daiichi-Sankyo Inc.

Quizartinib is currently under development for the treatment of patients 18 years of age or older with relapsed (including after HSCT) or refractory FLT3-ITD mutated AML, and has been granted Fast Track Status in the US and an Orphan Drug Indication in the United States, Europe and Asia.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following inclusion criteria prior to receive treatment:

1. Has provided written informed consent as approved per local regulations with privacy language in accordance with national regulations (eg, Health Insurance Portability and Accountability Act [HIPAA] authorization for US sites) prior to any protocol-related procedures
2. Is 18 years of age or the minimum legal adult age (whichever is greater) at the time of informed consent
3. Has morphologically documented primary AML or AML secondary to myelodysplastic syndrome (MDS) or other myeloproliferative neoplasms (MPN), as defined by the World Health Organization (WHO) 2008 classification with ≥5% blasts in bone marrow, with or without extramedullary disease
4. Is in relapse or refractory (R/R) to prior therapy, with or without HSCT

   1. Refractory is defined as:

      * participant did not achieve complete remission (CR), CR with incomplete platelet recovery (CRp), or CR with incomplete hematological recovery (CRi) under initial intensive therapy, or
      * did not achieve CR, CRp, CRi, or partial remission (PR) under initial sufficient time course of treatment with hypomethylating agents or low-dose cytarabine (LoDAC)
      * must have received at least one complete block of induction therapy seen as the optimum choice of therapy to induce remission or at least 4 cycles of therapy with a hypomethylating agent deemed sufficient to induce a response
   2. Relapse is defined as: relapse diagnosed by bone marrow assessment or by the appearance of peripheral blasts after the achievement of CR, CRp, or CRi, as defined by 2003 International Working Group criteria after AML therapy with or without consolidation or maintenance, and with or without HSCT
5. Has documented FLT3-ITD mutation in bone marrow or peripheral blood in relation R/R disease
6. Prior treatment with kinase inhibitors, including FLT3 targeted therapy or investigational FLT3 inhibitors is allowed
7. Has an Eastern Cooperative Oncology Group (ECOG) performance score 0-3
8. Discontinued prior AML treatment before the start of protocol treatment (except hydroxyurea or other treatment to control leukocytosis) for at least 2 weeks for cytotoxic agents, or for at least 5 half-lives for non-cytotoxic agents
9. Has creatinine clearance >25 mL/min, as calculated with the Cockcroft-Gault formula
10. Has serum potassium, magnesium, and calcium (serum calcium corrected for hypoalbuminemia) within institutional normal limits. Participants with electrolytes outside the normal range will be eligible if these values are corrected upon retesting following any necessary supplementation
11. Total serum bilirubin ≤1.5 × upper limit of normal (ULN)
12. Has serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 × ULN

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from enrollment:

1. Is eligible to enroll in a recruiting clinical trial of quizartinib or is currently enrolled in an ongoing clinical trial of quizartinib
2. Has previously participated in a randomized clinical study of quizartinib with an endpoint of survival that is not closed for efficacy
3. Has acute promyelocytic leukemia (AML subtype M3)
4. Has persistent, clinically significant ≥Grade 3 non-hematologic toxicity from prior AML therapy
5. Has clinically significant acute graft-versus-host disease (GvHD) or GVHD requiring initiation of treatment or treatment escalation within 21 days, and/or ≥Grade 3 persistent or clinically significant non-hematologic toxicity related to HSCT
6. Has uncontrolled or significant cardiovascular disease, including:

   * QTcF interval >450 ms
   * Bradycardia of less than 50 beats per minute (bpm) unless the patient has a pacemaker
   * Diagnosed or suspected long QT syndrome, or known family history of long QT syndrome
   * History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or torsade de pointes
   * History of second or third degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers, and have no history of fainting or clinically relevant arrhythmia with pacemakers.
   * Myocardial infarction within 6 months prior to screening
   * Uncontrolled angina pectoris within 6 months prior to Screening
   * New York Heart Association (NYHA) Class 3 or 4 congestive heart failure
   * Left ventricular ejection fraction (LVEF) ≤45% or institutional lower limit of normal
   * Uncontrolled hypertension
   * Complete left bundle branch block
7. Has active infection not well controlled by antibacterial, antifungal, and/or antiviral therapy
8. Has active hepatitis B or C, or other active clinically relevant liver disease
9. Is unwilling to receive infusion of blood products according to the protocol
10. Women are regarded as of childbearing potential if they are not post-menopausal (at least 2 years without menses) or surgically sterile (at least 1 month before enrollment).

    Highly effective contraception methods include: combined (estrogen and progestogen containing) hormonal methods associated with inhibition of ovulation, intra-uterine device; surgical sterilization (including bilateral tubal occlusion, partner's vasectomy) or sexual abstinence if this is the preferred and usual lifestyle of the participant
    1. If a heterosexually active woman of childbearing potential:

       * Either partner is unwilling or unable to use a highly effective contraceptive method (as described above) for the entire treatment period and for at least 6 months after the administration of the final dose of quizartinib
       * Is unwilling to refrain from donating or retrieving ova for her own use from the time of Screening and throughout the treatment period, and for 12 weeks after the administration of the final dose of quizartinib
       * Is pregnant - quizartinib should be permanently discontinued if pregnancy is confirmed
       * Is unwilling to refrain from breastfeeding from the time of Screening and throughout the protocol period, and for 25 days after the administration of the final dose of quizartinib
    2. If a man whose sexual partner is a woman of childbearing potential:

       * Either partner is unwilling or unable to use a highly effective contraceptive method (as described above) for the entire treatment period and for at least 6 months after completion of protocol treatment
       * Is unwilling to refrain from freezing or donating sperm starting at Screening and throughout the treatment period and 105 days after the administration of the final dose of quizartinib
11. Has any medical condition, serious intercurrent illness, or other circumstance that, in the treating physician's judgment, could jeopardize the participant's safety

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult